CLINICAL TRIAL: NCT01897051
Title: Hemodynamic Response of Rifaximin and Non-selective β-blocker Combination Therapy Versus Non-selective β-blocker Monotherapy in Cirrhotic Patients With Esophageal Varices
Brief Title: Rifaximin and Propranolol Combination Therapy Versus Propranolol Monotherapy in Cirrhotic Patients
Acronym: RECOVER
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Moon Young Kim, Associate Professor, Divistion of Gastroenterology and Hepatology, Department of Internal Medicine, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR310037
Record Dates: First submitted 2013-07-01; First posted 2013-07-11 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Liver Cirrhosis; Portal Hypertension
Keywords: Liver cirrhosis; Portal hypertension; Hepatic Venous Pressure Gradient; Rifaximin
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal | interventions — Rifaximin; Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination therapy (Experimental): Rifaximin(normix®)+nonselective beta-blocker(Propranolol)
  Interventions: Drug: Rifaximin + propranolol
- Monotherapy (Placebo Comparator): nonselective beta-blocker(Propranolol) + Placebo(of Rifaximin)
  Interventions: Drug: Propranolol + Placebo

INTERVENTIONS:
Drug: Rifaximin + propranolol — 1. Rifaximin : taking 400mg three times a day in the study period (total 1,200 mg per day)
  2. Propranolol : taking 40mg twice a day to start. If patient is tolerable and systolic blood pressure is above 90 mmHg, the dosage can be increased by doubling to every other day upto the 360mg per day.
  (Target heart rate : 25% reduction in baseline heart rate or at least 55 times per minute).
  If patient is not tolerable, we can reduce the dosage step-by-step until the adverse symptoms is disappeared.
  Other Names: Normix; Propranolol
  Arms: Combination therapy
Drug: Propranolol + Placebo — 1. Placebo of Rifaximin : taking 400mg three times a day in the study period (total 1,200 mg per day)
  2. Propranolol : taking 40mg twice a day to start. If patient is tolerable and systolic blood pressure is above 90 mmHg, the dosage can be increased by doubling to every other day upto the 360mg per day.
  (Target heart rate : 25% reduction in baseline heart rate or at least 55 times per minute).
  If patient is not tolerable, we can reduce the dosage step-by-step until the adverse symptoms is disappeared.
  Other Names: Non-selective beta-blocker; Placebo of Rifaximin
  Arms: Monotherapy

SUMMARY:
To reduce portal pressure, the only recommended medication is nonselective beta blocker(NSBB). However, NSBB has some limitation to apply clinically because of poor response rate and compliance.

Recent literature has supported the role of bacterial translocation as a mediator of splanchnic vasodilatation and portal hypertension. This stimulates the release of pro-inflammatory cytokines and the activation of the vasodilator NO resulting in a more pronounced deterioration of the baseline hyperdynamic circulatory state. Selective gut decontamination with Rifaximin can induce inhibition of bacterial translocation and associated worsening of portal hypertension. The investigators hypothesized that Rifaximin plus NSBB could result in decrease of portal pressure in cirrhotic patients with esophageal varices.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis:diagnosed based on histology or unequivocal clinical, sonographic, and laboratory findings
* 19≤age≤75
* Hepatic venous pressure gradient > 12 mmHg
* Informed consent

Exclusion Criteria:

* Shock status requiring vasopressor
* Active infection, for example Spontaneous bacterial peritonitis
* Acute renal failure patients of any cause
* Clinically relevant coronary artery disease(NYHA functional angina classification III/IV),congestive heart failure NYHA III/IV), clinically relevant cardiomyopathy, history of myocardial infarction in the past 12 months
* Poorly controlled hypertension (BP 150/100mmHg)
* Hepatocellular carcinoma
* History of another primary malignancy ≤ 3years
* Medical or psychological conditions that would not permit the subject to complete thte study or sign informed consent
* Pregnancy or lactation period
* Serum creatinine ≧ 6mg/dL
* Involvement in the conduct of other study within 30 days
* Known hypersensitivity to Rifaximin or propranolol
* Dysarrhythmia, inappropriate for study on investigator's judgment

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2013-07; Primary Completion 2017-02 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Hepatic vein pressure gradient(HVPG) | Change from baseline heptic vein pressure gradient at 6 weeks
  After measurement of baseline HVPG, patients will be randomized to treatment group of Rifaximin + Propranolol or Propranolol + Placebo. And 6 weeks after treatment, follow-up measurement of HVPG will be performed to evaluate efficacy of two regimens

SECONDARY OUTCOMES:
occurence of gastrointestinal bleeding | upto 6 months after initiation of treatment
  when gastrointestinal bleeding occurs, after initiation of treatment, endoscopy will be performed to evaluate status of bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Moon Young Kim, MD,PhD, Principal Investigator — Yonsei University; Moon Young Kim, M.D., PhD., Study Chair — Yonsei University Wonhu College of Medicine Wonju Severance Christian Hospital
Locations (2):
- South Korea (2):
  - Yonsei University Wonju Severance Cristian Hospital, Wŏnju, Gangwon-do
  - Wonju Severance Christian Hospital, Wŏnju

REFERENCES:
- [Background] Rasaratnam B, Kaye D, Jennings G, Dudley F, Chin-Dusting J. The effect of selective intestinal decontamination on the hyperdynamic circulatory state in cirrhosis. A randomized trial. Ann Intern Med. 2003 Aug 5;139(3):186-93. doi: 10.7326/0003-4819-139-3-200308050-00008. PMID 12899586
- [Background] Vlachogiannakos J, Saveriadis AS, Viazis N, Theodoropoulos I, Foudoulis K, Manolakopoulos S, Raptis S, Karamanolis DG. Intestinal decontamination improves liver haemodynamics in patients with alcohol-related decompensated cirrhosis. Aliment Pharmacol Ther. 2009 May 1;29(9):992-9. doi: 10.1111/j.1365-2036.2009.03958.x. Epub 2009 Feb 7. PMID 19210289
- [Background] Gonzalez A, Augustin S, Perez M, Dot J, Saperas E, Tomasello A, Segarra A, Armengol JR, Malagelada JR, Esteban R, Guardia J, Genesca J. Hemodynamic response-guided therapy for prevention of variceal rebleeding: an uncontrolled pilot study. Hepatology. 2006 Oct;44(4):806-12. doi: 10.1002/hep.21343. PMID 17006916
- [Background] Ripoll C, Banares R, Rincon D, Catalina MV, Lo Iacono O, Salcedo M, Clemente G, Nunez O, Matilla A, Molinero LM. Influence of hepatic venous pressure gradient on the prediction of survival of patients with cirrhosis in the MELD Era. Hepatology. 2005 Oct;42(4):793-801. doi: 10.1002/hep.20871. PMID 16175621
- [Background] Kumar M, Kumar A, Hissar S, Jain P, Rastogi A, Kumar D, Sakhuja P, Sarin SK. Hepatic venous pressure gradient as a predictor of fibrosis in chronic liver disease because of hepatitis B virus. Liver Int. 2008 May;28(5):690-8. doi: 10.1111/j.1478-3231.2008.01711.x. PMID 18433395